CLINICAL TRIAL: NCT06427967
Title: Beyond Watching and Waiting: A Pilot Study of a Novel Social Emotional Learning Curriculum-Based Intervention Designed for Youth With Epilepsy at Increased Risk of Future Mental Illness
Brief Title: A Novel Social Emotional Learning Curriculum for Youth With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Charles H. Hood Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-43875; 4301210001 (Other Grant/Funding Number: Charles F. Hood Foundation)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy
Keywords: Youth with epilepsy (YWE); Positive Youth Development; Social-Emotional Learning; Social Ecological Model; Youth Thrive Framework; Perceived Social Support; Health-Related Quality of Life; Adult Epilepsy Self-Management Measurement Instrument
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: One-group pretest-posttest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Novel Social-Emotional Learning (SEL) curriculum (Experimental): Participants assigned to this arm will receive Project Dream Team, the new 5 session SEL curriculum for YWE.
  Interventions: Behavioral: Project Dream Team

INTERVENTIONS:
Behavioral: Project Dream Team — Five total sessions, 60-minutes each, with one session every 7 days (+/- 21 days between sessions), Session activities include discussion prompts, interactive learning methods, skill rehearsals, mindfulness / somatic exercises and lecture slides facilitated by a trained facilitator.

SUMMARY:
Youth with epilepsy (YWE) are significantly more likely than their peers without epilepsy to experience isolation, interpersonal victimization, and low relationship satisfaction. This is a serious health concern. Poor social support, real or perceived, is consistently correlated to worsened outcomes in every domain of health-related quality of life. As YWE are two to five times more likely than their peers without epilepsy to develop a mental health condition, poor social support is likely a bidirectional risk factor.

Currently, there are no best practices or recommendations for clinicians or other youth-serving professionals to reference when it comes to improving the perceived social support of YWE specifically.

The research team has drawn from multiple fields of scientific knowledge to develop a novel intervention that aims to provide YWE with knowledge, skills, connections, and positive emotional support that can help them to bolster their support system at every level of the social ecological model (SEM). The proposed study is a pilot of this intervention to test its acceptability and appropriateness according to YWE participants ages 12 to 26. The intervention's impact on participants social-emotional learning skills and the feasibility of expanding the study protocol for use in a large, multisite randomized control trial will also be explored.

The goal of this research study is to help evaluate a new program for young people diagnosed with epilepsy that will build up young people's social opportunities, interpersonal skills, and sources of emotional support. The investigators want to research the impact of this program. From this study, the investigators hope to learn what the program does well, and in what ways it could be improved from the perspective of YWE.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, and communicate in English at 3rd grade level
* Active epilepsy diagnosis (currently on anti-seizure medication or does not yet meet remission standards of 10 years without seizure and off all medication)
* Epilepsy diagnosis clinically established for at least 6 months prior to the time of recruitment
* The pediatric neurologist feels the patient would benefit from program participation.
* Able to consistently join meetings on Zoom with functional audio and video reception

Exclusion Criteria:

* During the consent process, if an eligible potential participant feels that participation would pose too much of a burden on their health or mental wellbeing, they will be excluded.

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of study processes | 4 months
  Number of sessions attended per participant.
Acceptability of the intervention | 4 months
  A likert scale will be used to assess satisfaction from 1 to 10 where 10 is highly acceptable and 1 is not acceptable.

SECONDARY OUTCOMES:
Change in perceived social support (PSS) | Baseline, 4 months
  This outcome will be assessed with the Youth Thrive (YT) Framework Survey Part 1: Social Connections and Concrete Supports combine subscales. Each YT subscale includes 10 to 16 individual Likert scale questions. Scores are generated by assigning values of 1 to 5 to the Likert scale (1 = not at all like me, 5 = very much like me) for 'positive items' and an inverse value scale for 'negative items' and then totalling all the items within the subscale. Higher total scores indicate a higher level of PSS.

OTHER OUTCOMES:
Change in social emotional skills and behaviors | Baseline, 4 months
  The Youth Thrive (YT) Framework Survey Part 2: Youth Resilience, Cognitive and Social-Emotional Competence subscales will be used to assess this outcome. Each YT subscale includes 10 to 16 individual Likert scale questions. Scores are generated by assigning values of 1 to 5 to the Likert scale (1 = not at all like me, 5 = very much like me) for 'positive items' and an inverse value scale for 'negative items' and then totalling all the items within the subscale. Higher total scores indicate a greater depth of knowledge, higher mastery over key skills and more frequent use of prosocial behaviors.
Change in leveraging social support for epilepsy self management | Baseline, 4 months
  This outcome will be assessed using the 25 subscale items from the Adult Epilepsy Self-Management Measurement Instrument (AESMMI-65). The responses are Likert scale-rated from 0 to 5 for positively phrased items, and inversely scored for negatively phrased items. Each subscale will be scored individually and also totaled for a single composite score. Higher scores indicate higher use of effective epilepsy self-management strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Douglass, MD, Principal Investigator — Boston Medical Center, Department of Neurology
Locations (1):
- Boston Medical Center, Neurology and remote, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No